CLINICAL TRIAL: NCT05471492
Title: A PHASE 2A, MULTICENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY WITH AN OPEN LABEL CHRONIC TREATMENT PERIOD TO EVALUATE THE EFFICACY, SAFETY, AND PHARMACOKINETICS OF PF-06480605 IN ADULT PARTICIPANTS WITH MODERATE TO SEVERE CROHN'S DISEASE
Brief Title: Study to Evaluate the Efficacy and Safety of PF-06480605 in Adult Participants With Moderate to Severe Crohn's Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial not started; change in Sponsor, a new trial to be registered by the new Sponsor
Sponsor: Telavant, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7541009; 2022-001259-18 (EudraCT Number)
Record Dates: First submitted 2022-07-18; First posted 2022-07-22 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Crohn Disease
Keywords: Crohn Disease, PF-06480605, SES-CD, CDAI,
MeSH Terms: conditions — Crohn Disease; Anemia, Dyserythropoietic, Congenital

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group 1 (Experimental): PF-06480605 150 mg
  Interventions: Drug: Investigational Product
- Treatment Group 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Investigational Product — PF-06480605 150 mg
  Arms: Treatment Group 1
Drug: Placebo — Placebo
  Arms: Treatment Group 2

SUMMARY:
This Phase 2a, multicenter, randomized, double-blind, placebo-controlled study examines subcutaneous dose of PF-06480605 150 mg administered every 4 weeks in participants with moderate to severe active Crohn's Disease to characterize safety, efficacy, pharmacokinetics, and immunogenicity

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of ileocolonic or colonic CD with at least 3 months or longer prior to the baseline;
* Central read total SES-CD score of ≥7. For isolated ileal disease, SES-CD total score should be ≥4;
* An average daily liquid/very soft SF ≥4 or daily AP score ≥2.0;
* CDAI between 220 and 450 inclusive;
* Must have inadequate response to, loss of response to, or intolerance to at least one conventional therapy for CD

Exclusion Criteria:

* Diagnosis of indeterminate colitis, microscopic colitis, ischemic colitis, infectious colitis, radiation colitis, diverticular disease, UC, or clinical findings suggestive of UC;
* Presence of active (draining) fistulae or intra-abdominal or perineal abscesses;
* Strictures or stenosis with obstructive symptoms;
* Short bowel syndrome;
* History of bowel perforation requiring surgical intervention within the past 12 months prior to baseline;
* Previous bowel surgery resulting in an existing stoma. Participants who have a j-pouch are excluded, as a j-pouch can result in a stoma;
* History of bowel surgery within 6 months prior to baseline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with endoscopic response 50 | Week 14
  Endoscopy response 50 (SES-CD50) is defined as a reduction from baseline in Simple Endoscopic Score for Crohn's Disease (SES-CD) at least 50% or more. SES-CD score assesses the presence of ulcers, the percentage of ulcerated surface, the percentage of affected surface, and the presence of narrowing using scales ranging from 0 to 3 in each following bowel segment: Ileum, right colon, transverse colon, left colon, rectum. The score ranges from 0 to 60 with higher score indicating more severe disease.

SECONDARY OUTCOMES:
Proportion of participants with a Crohn's Disease Activity Index (CDAI) clinical remission | Week 14
  Clinical remission is defined as CDAI < 150. CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid stools, extent of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity.
Proportion of participants achieving endoscopic remission | Week 14
  Endoscopic remission is defined as SES-CD < 4 and at least 2-point reduction versus Baseline and no individual subscore > 1
Proportion of participants achieving endoscopic mucosal healing | Week 14
  Endoscopic mucosal healing defined as complete absence of ulcers in SES-CD
The proportion of participants with Inflammatory Bowel Disease Questioners (IBDQ) total score ≥170 | Week 14
  Inflammatory Bowel Disease Questionnaire (IBDQ) score ranges from 32 to 224. A higher score indicates better quality of life. A score of at least 170 corresponds to clinical remission.
Proportion of participants achieving endoscopic response | Week 52
  Endoscopic response defined as improvement of SES-CD score at least 50% from baseline
Proportion of participants with a CDAI clinical remission | Week 52
  Clinical remission is defined as CDAI < 150. CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid stools, extent of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity.
Proportion of participants achieving endoscopic remission | Week 52
  Endoscopic remission is defined as SES-CD < 4 and at least 2-point reduction versus Baseline and no individual subscore > 1
Proportion of participants achieving endoscopic mucosal healing | Week 52
  Endoscopic mucosal healing defined as complete absence of ulcers in SES-CD
Proportion of participants with a CDAI clinical remission | up to week 52
  CDAI < 150 overtime during induction treatment period
Proportion of participants with a CDAI clinical response | Up to week 52
  As defined by a decrease from baseline in CDAI score of at least 100 points or more
Proportion of participants achieving Patient Reported Outcome 2 (PRO2) clinical response | Up to week 52
  PRO2 clinical response is define by improvement in number of liquid/soft stool frequency and abdominal pain score at least 30% from baseline
Proportion of participants achieving PRO2 clinical remission | Up to week 52
  PRO2 clinical remission is defined as SF≤2.5 and AP≤1
Incidence of AEs or SAEs including events leading to withdrawal due to abnormalities in laboratory, vital signs, and ECG. | up to week 52
Incidence of development of severe and serious infections | Up to week 52

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7541009